CLINICAL TRIAL: NCT01410136
Title: A Post Market Study to Evaluate the Chondrofix® Osteochondral Allograft Utilized for Treatment of Subjects With Cartilage Lesions in the Knee
Brief Title: Chondrofix Osteochondral Allograft Prospective Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment and decreased need for clinical data to support product
Sponsor: Zimmer Orthobiologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSU2010-14B
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Articular Cartilage Disorder; Degeneration; Articular Cartilage; Chronic Cartilage Injury; Acute Cartilage Injury; Defect of Articular Cartilage
Keywords: Knee; Femur; Articular cartilage; Lesions; Defects; Osteochondral graft; Cartilage treatments; Osteochondritis Dissecans; OCD
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chondrofix (Other): Subjects with one or two confirmed knee articular cartilage lesion(s) each less than 8cm2, of the femoral condyle or trochlear groove
  Interventions: Procedure: Chondrofix Osteochondral Allograft

INTERVENTIONS:
Procedure: Chondrofix Osteochondral Allograft — Allogeneic, cylindrical, decellularized, osteochondral graft composed of hyaline cartilage and bone
  Other Names: Chondrofix

SUMMARY:
The overall study objective is to evaluate Chondrofix Osteochondral Allograft ("Chondrofix") for the repair of osteochondral lesions in the knee. This includes, but is not limited to primary cartilage lesion repair and revision of failed prior cartilage repair treatments. The study hypothesis is that Chondrofix Allograft will provide pain relief and functional improvement as demonstrated by a comparative analysis of baseline clinical evaluations at 24 months of follow-up.

DETAILED DESCRIPTION:
Knee cartilage injuries are a major cause of pain and functional impairment in young to middle age adults and can lead to progressive joint degeneration. In response to challenges with current cartilage repair options, Chondrofix Allograft was developed as an off-the-shelf treatment option adding to the variety of cartilage reparation offerings.

This study is a multicenter, prospective, post-market clinical outcomes study designed to assess the clinical outcomes of Chondrofix Allograft used in the treatment of both primary and revision cartilage repair cases. Study design includes up to 6 qualified investigational sites with 50 subjects enrolled across all centers during an 18 month enrollment period. Study subjects will be followed postoperatively for 5 years. The Investigators who are responsible for the conduct of this study in compliance with this protocol will be orthopedic surgeons who are skilled in the techniques of articular cartilage repair.

ELIGIBILITY:
Inclusion Criteria:

Generally, the following inclusion criteria must be met, however, this is not a complete list.

* Male and non-pregnant female subjects between 18 and 70 years; subject must be skeletally mature
* If female, subjects are not pregnant at time of surgery and do not plan on becoming pregnant during the first 24 months of the study
* Up to two (2) cartilage lesion(s), each measuring less than 8 cm2, of the femoral condyle or trochlear groove of the knee
* Localized knee pain unresponsive to conservative treatment (e.g., medication, bracing, physical therapy) and/or previous surgical intervention

Exclusion Criteria:

Generally, if a potential participant meets any of the following criteria, they will not be eligible for this study. Additionally, more criteria will be evaluated to confirm eligibility as this list is not a complete list of criteria.

* Concurrent participation in another clinical trial
* Cartilage lesion location is such that the implanted graft(s) will not be adequately shouldered
* Bipolar articular cartilage involvement (or kissing lesions) of the ipsilateral compartment (i.e., > than ICRS Grade 2 on the opposing articular surface)
* Is receiving pain medication other than NSAIDs or acetaminophen for conditions unrelated to the index knee condition
* Subject had any other cartilage repair procedure other than debridement performed in conjunction with or 6 months prior to implantation of a Chondrofix Osteochondral Allograft
* Prior or concurrent total meniscectomy of the index knee
* Uncorrected mal-alignment of the index knee
* Have smoked or used nicotine products within the past 6 months
* Body Mass Index > 35 (BMI=kg/m2)
* Has any contraindications for MRI
* Requires any of the following concomitant procedures performed in conjunction with or has had performed within 6 months prior to implantation of a Chondrofix Allograft: distal realignment, high tibial osteotomy, ligament reconstruction, and/or patellar realignment procedure
* Septic or reactive arthritis or systemic disease (e.g., rheumatoid arthritis, gout or prior history of gout or pseudo gout)
* Sickle cell disease, hemochromatosis, or autoimmune disease
* Unstable cardiovascular, renal, hepatic, endocrine and/or pulmonary disease, cancer or uncontrolled diabetes
* HIV or other immune-deficient state including subject on immunosuppressant therapies
* Deficiency limiting ability to perform an objective functional assessment of the operative knee or an inability to adhere to a post-operative rehabilitation protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
KOOS Subscale | 24 Months
  The overall mean change from baseline to 24 months in the KOOS Pain and KOOS Function in Daily Living (ADL) subscale scores.

SECONDARY OUTCOMES:
X-ray & MRI Evaluation | Baseline and 1.5, 3, 6, 12, 24, & 60 months
IKDC Knee Examination | Baseline & 1.5, 3, 6, 12, 24, & 60 months
Subject Reported Questionnaires | Baseline and 1.5, 3, 6, 12, 24, 36, 48, and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Nikesha N Harrington, Study Chair — Zimmer Orthobiologics, Inc.
Locations (5):
- United States (5):
  - Plancher Orthopaedics and Sports Medicine, Cos Cob, Connecticut
  - The Orthopaedic Group, LLC, New Haven, Connecticut
  - Orthopaedic Research Foundation, Inc., Greenwood, Indiana
  - Cartilage Repair Center, Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Specialized Orthopaedics and Sports Medicine, Columbus, Ohio